CLINICAL TRIAL: NCT01361425
Title: Effectiveness Of Anti-Hypertensive Treatment In Stable Pregnant Women With Severe Pre-Eclampsia: Randomized Placebo-Controlled Clinical Trial
Brief Title: Anti-Hypertensive Treatment In Stable Pregnant Women With Severe Pre-Eclampsia (Metildopape)
Acronym: METILDOPAPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: M.D; M.S Carlos Noronha Neto, IMIP
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: METILDOPA PE 1
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-04

CONDITIONS: Preeclampsia
Keywords: hypertension; ultrasonography; preeclampsia; clinical trials; treatment; methyldopa
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Methyldopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methildopa (Experimental): pregnant women with stable severe pre-eclampsia will use methildopa (1,5g/day)
  Interventions: Drug: methildopa
- placebo (Placebo Comparator): stable pregnant women with severe preeclampsia will use placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methildopa — methildopa, 1,5g/day (500mg 8/8 hours, orally)
  Other Names: ALDOMET
  Arms: methildopa
Drug: placebo — placebo 500mg 8/8h, orally
  Other Names: Placebo comparator
  Arms: placebo

SUMMARY:
Introduction: Hypertensive emergency in pregnant women with pre-eclampsia should be treated for preventing stroke and placental abruption. However, the benefit of antihypertensive medication maintenance remains unclear, mainly due to the potential risk of fetal growth restriction.

DETAILED DESCRIPTION:
Objectives: To evaluate the effectiveness of antihypertensive treatment maintenance with 1.5 g / day of methyldopa for controlling maternal blood pressure in pregnant women with severe pre-eclampsia and stable blood pressure. Methods: A clinical, randomized, triple-masked, placebo-controlled study will be conducted at the Instituto de Medicina Integral Prof. Fernando Figueira from March 2011 to March 2012. The study will include 200 patients with severe preeclampsia between 20 to 34 weeks of gestation, which will be randomized into two groups: placebo and methyldopa. Patients with more severe hypertensive disorders, congenital anomalies and maternal medical complications or conditions that may compromise the mother-child well-being will be excluded from the study. The primary outcomes will be: systolic, diastolic and mean maternal heart rate, need for association with another antihypertensive agent, need and reason for discontinuation of treatment, frequency of hypertensive peaks and uncontrolled hypertension. The variables relating to maternal characteristics of pregnancy, clinical and obstetric complications during pregnancy and after delivery, and adverse perinatal outcomes will be considered secondary outcomes. After inclusion of patients in the study, numbered boxes containing methyldopa or placebo will be offered to patients with appropriate explanations about oral administration. The initial dose of methyldopa is 1.5 g / day divided into three daily doses and can be reduced to 1.0 g / day or increased to 2.0 g / day depending on the clinical need of patients. On the other group, three tablets / day of placebo will be administered and this dose may be reduced or increased to two tablets to four tablets per day. Statistical analysis will be performed using the statistical program Epi-Info 3.5.1. and Minitab, version 14.2. for Windows. The analysis will be performed with the groups identified as A or B, and the secrecy will be broken only after obtaining the results and preparing the tables or by resolution of the Committee for External Monitoring. Categorical variables will be compared in contingency tables, using chi-square and Fisher exact test, when appropriate. Risk ratio (RR) and its 95% confidence interval will be calculated as a measure of relative risk. Regarding the quantitative variables, if they have normal distribution, comparison between groups will be performed using the Student t test for unpaired samples. If it is found that the distribution is not normal, the nonparametric Mann-Whitney test will be used.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancy
* severe preeclampsia
* life fetus
* stable blood pressure
* gestational age between 20 weeks and 34 weeks

Exclusion Criteria:

* fetal anomalies
* antihypertensive drugs use
* others drugs use
* active labour
* tabagism
* Intra-Uterine Growth Restriction process

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Arterial blood pressure stabilization after methildopa use | one week
  Stabilization of arterial blood pressure in stable pregnant women with severe pre-eclampsia after methildpa or placebo use will be investigated, as well as occurrence of complications for mother and fetus.

SECONDARY OUTCOMES:
Complications in stable pregnant women with severe preeclampsia after methildopa use | one week
  Complications in stable pregnant women with severe preeclampsia after methildopa use

CONTACTS AND LOCATIONS:
Overall Officials: Melania M Amorim, PHD, Study Director — Fernando Figueira IMIP
Locations (2):
- Brazil (2):
  - Melania Maria Ramos de Amorim, Campina Grande, João Pessoa
  - Leila Katz, Recife, Pernambuco